CLINICAL TRIAL: NCT04195997
Title: Multi-center Application of Bivalirudin in High-risk Bleeding Patients With Non-valvular Atrial Fibrillation Undergoing Percutaneous Left Atrial Appendage Occlusion
Brief Title: Multi-center Application of Bivalirudin in Left Atrial Appendage Occlusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZS-2018-81
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Evaluate the Safety and Efficacy of Bivalirudin in Decreasing Bleeding Risk
MeSH Terms: interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- bivalurudin (Experimental): Bivalirudin will be given as a bolus of 0.75 mg/kg once transseptal puncture is successully performed with no pericardial effusion. An additional bivalirudin bolus of 0.3 mg/kg was given if the activated clotting time 5 minutes after the initial bolus was less than 225 seconds.
  Interventions: Drug: Bivalirudin
- heparin (Active Comparator): Heparin will be administered at a dose of 70 to 100 units per kilogram in patients not receiving glycoprotein IIb/IIIa inhibitors. Subsequent adjustment of the heparin dose on the basis of the activated clotting time will be left to the discretion of the treating physicians.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin — Patients would be given anticoagulant therapy with bivalirudin in left atrial appendage occusion.
  Arms: bivalurudin
Drug: Heparin — heparin during left atrial appendage occlusion.
  Arms: heparin

SUMMARY:
The study is an investigator-sponsored, prospective, multicenter, randomized, open-label study designed to compare efficacy and safety between bivalirudin and heparin in patients with non-valvular atrial fibrillation undergoing percutaneous left atrial appendage occlusion.

DETAILED DESCRIPTION:
Bivalirudin, a direct thrombin inhibitor, emerged as an important representative of intravenous anticoagulant and has been recommended for treatment of acute coronary syndromes with percutaneous coronary intervention according to American and European guidelines.On concerns of risk of bleeding and thrombosis,bivalirudin shows significant advantages over traditional glycoprotein inhibitors(GPI).However,the research about the application of bivalirudin for patients at high-risk of stroke and bleeding with non-valvular atrial fibrillation is still at blank stage.Percutaneous left atrial appendage occlusion is nowadays an effective alternative for stroke prevention and its targeted population is featured as CHA2DS2 score≥2 and/or HAS-BLED score≥3.The purpose of this multi-center trial is to evaluate the safety and peri-procedual efficacy of bivalirudin for patients at high-risk atrial fibrillation patients undergoing percutaneous left atrial appendage occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 60 years;
2. non-valvular atrial fibrillation patients with contraindication for long-term oral anticoagulant or occurrence or stroke in spite of regular administration of medication;
3. CHA2DS2 score≥2 and/or HAS-BLED score≥3;
4. Provide written informed consent.

Exclusion Criteria:

1. Left atrial diameter≥65mm;Severe mitral regurgitation；percardial effusion>3mm；LVEF<35%;
2. Peri-procedual thrombus in left atrial and/or left atrial appendage confirmed by TEE;
3. Other comorbidities requiring for use of anticoagulants.
4. Life expectancy ≥ 1 year;
5. CHA2DS2 score ≤1 and HAS-BLED score≤2;
6. Active bleeding or bleeding constitution, bleeding tendency, including GI or urinary tract hemorrhage (3 months), cerebral hemorrhage (6 months) or cerebral infarction history (3 months), etc;
7. Other disease may lead to vascular lesions and secondary bleeding factors (such as active gastric ulcer, active ulcerative colitis, intra-cerebral mass, aneurysm, etc.);
8. Severe renal insufficiency (eGFR < 30 mL/min/ 1.73 m2); Elevated AST, ALT level higher than three times of the normal upper limit; Advanced heart failure (NYHA classification grading of cardiac function ≥ Ⅲ) Complicated with immune system diseases；
9. Abnormal hematopoietic system：platelet count < 100 * 109 / L or > 700 * 109 / L，white blood cell count < 3 * 109/L etc;
10. Suffering from acute infections ,infectious diseases or other serious diseases, such as malignant tumors;
11. Known intolerance, or contraindication to any antithrombotic medication Known allergy to the study drugs and instruments (UFH, bivalirudin, aspirin and clopidogrel, stainless steel, contrast agents, etc.), or those allergic constitution.

    Non-cardiac co-morbid conditions are present that may result in protocol non-compliance;
12. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period;
13. Patient's inability to fully cooperate with the study protocol

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 7 days
  a composite of all cause death, stroke
Major bleeding | 7 days
  BARC types 2-5 bleeding;TIMI major bleeding or GUSTO moderate to severe bleeding

SECONDARY OUTCOMES:
Creatine kinase-MB increase | up to postprocedural 72 hours
  creatine kinase-MB increase >3 times upper limit of normal
Major bleeding | 60 days
  BARC types 2-5 bleeding;TIMI major bleeding or GUSTO moderate to severe bleeding
Major adverse cardiac events | 60 days
  a composite of all cause death, stroke，heart failure
Device-related thrombus | 60 days
  rate of stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: XIAOCHUN ZHANG, MD, Principal Investigator — Department of Cardiology, Zhongshan Hospital, Fudan University
Locations (1):
- Zhongshan Hopital of Fudan University, Shanghai, Shanghai Municipality, China